CLINICAL TRIAL: NCT05938114
Title: Effectiveness of Two Bone Substitutes, Natural and Synthetic, in Preserving the Alveolar Ridge of Single-rooted Teeth: a Pilot Single-blind, Parallel Randomised Controlled Trial
Brief Title: Comparison of the Use of Natural and Synthetic Bone Substitutes in Dental Implants
Acronym: BSNS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Central Lancashire (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Principal Investigator, Fadi Barrak, Course Lead and Senior Lecturer, University of Central Lancashire, School of Dentistry, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HEALTH 01032; IRAS ID: 316275 (Other: NHS Health Research Authority)
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Alveolar Ridge Augmentation
Keywords: Ridge Preservation; Bone Substitutes; Alveolar Bone
MeSH Terms: interventions — Bio-Oss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Bonalive®) (Experimental): The test bone substitute is Bonalive®, bioactive glass S53P4, which contains SiO2, Na2O, CaO, and P2O5 (granule size 0.5-0.8mm). Bonalive® is osteoconductive, meaning that it has the ability of promoting bone growth across the granules and the grafting area and slowly replace it with new bone over time. Bonalive® is osteostimulative and has antibacterial properties
  Interventions: Other: Bonalive
- Group B ( Bio-Oss®) (Active Comparator): The comparator is Bio-Oss®, deproteinized bovine bone granules (granule size 0.25- 1mm). Bio-Oss® is osteoconductive, which means it acts as a scaffold only for new bone to grow.
  Interventions: Other: Bio-Oss®

INTERVENTIONS:
Other: Bonalive — Bonalive® is a bioactive glass synthetic bone substitute material that has been shown to have a low substitution rate and antibacterial properties. It has been used successfully in the orthopaedics, craniofacial and ear nose and throat (ENT) specialities for the treatment of osteomyelitis, sinusitis and bony cyst cavities. There have also been a few maxillofacial surgery case reports on its usage in the jaws.
  Arms: Group A (Bonalive®)
Other: Bio-Oss® — Bio-Oss® is a bovine xenogeneic bone graft substitute that is widely used in regenerative dentistry. Bio-Oss® is very similar to human bone in its structure and chemical make-up. The material's porosity allows for vascularisation and new bone formation.
  Arms: Group B ( Bio-Oss®)

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of a natural and synthetic bone substitute in preserving the alveolar ridge (bone) of a single- rooted tooth after an extraction.

The main question it aims to answer:

Is there a difference between natural (Bio-Oss®) and synthetic (Bonalive®) bone substitutes in preserving the alveolar ridge dimensions based on changes in the width of the alveolar ridge (expressed in millimetres) from augmentation (baseline) to 24-week follow-up (post augmentation)?

Participants will have a tooth extraction and a bone substitute will be inserted into their socket immediately after. Participants will be divided into two equal groups and those in group A will receive Bio-Oss® while those in group B will receive Bonalive®. In both groups measurements of the alveolar bone will be taken when the bone substitute is inserted and 24 weeks after the insertion of the bone substitute. These measurements will be used to compare the effectiveness of Bio-Oss® and Bonalive in preserving the alveolar bone of a tooth after an extraction.

DETAILED DESCRIPTION:
It is a pilot single-blind two-arm parallel randomised control trial that aims to assess the differences between two bone substitutes, natural versus synthetic. The study will mimic the routine practice, and patients will be randomly allocated to receive either natural (control) or synthetic (intervention) bone substitutes. The patient follow-up period will be 24 weeks from the baseline data collection point.

The University of Central Lancashire will lead the study in collaboration with Imperial College London and dental clinics in Midlands, Southeast and Northwest England. We will recruit 34 patients who require tooth extractions and divide them into two equal groups. Patients in group A will receive Bio-Oss® , while those in group B will receive Bonalive® For both groups, the bone substitute will be inserted immediately after an extraction, and the socket will be sealed with a membrane sutured in place. Patients in both groups will be reviewed after 2 weeks to remove the suture. Patients will have another review at 24 weeks, during which the researcher will take a scan or mould, a photograph, and a small biopsy sample of the area where the bone substitute was placed. Measurements obtained at the 24-week follow-up will be used to evaluate the effectiveness and differences between natural and synthetic bone substitutes in preserving the bone supporting a tooth after an extraction.

The results of this pilot study will inform the design and implementation of a full-scale randomised controlled trial to investigate the effectiveness of bioactive glass-derived bone compared with bovine-derived bone in preserving the alveolar bone of a tooth after an extraction

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18) in need of extraction of a single-rooted tooth attending the clinics selected for the study
* Single units in a dentate patient
* Non-surgical extraction - no flap raised, and no bone removed Intact socket walls post-extraction
* Bleeding sockets
* Stable periodontal health

Exclusion Criteria:

* Multiple adjacent extractions
* Presence of active periodontal disease
* Socket walls not intact - >50% bone loss in any of the four walls
* Sclerotic sockets post-extraction - the socket does not fill up with blood post-extraction
* Denture wearer - the extraction socket site under the load of a denture
* Patients on medication that can affect bone healing e.g., bisphosphonates (oral or intravenous), selective serotonin reuptake inhibitors (SSRI), methotrexate, proton pump inhibitors (PPI)
* Uncontrolled diabetes Smokers Immunosuppressed Patients
* Patients with a history of myocardial Infarction in the last year ASA Class > II patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure is the change in the width of the alveolar ridge | Outcome data will be collected at baseline and week 24
  The change in the width of the alveolar ridge is expressed in millimetres and it will be obtained using intra-oral scanners (this does not involve radiographs) or impressions and clinical photographs.

SECONDARY OUTCOMES:
Change in height of the alveolar bone. | This outcome data will be collected at baseline and at week 24
  The change in height of the alveolar bone expressed in millimetres. Assessment will be done using the periapical radiographs taken pre-extraction and at 24-week follow-up and intra-oral scanners (this does not involve radiographs) or impressions and clinical photographs.
Changes in the vertical crestal bone level | This outcome data will be collected at baseline and at week 24
  The change in the vertical crestal bone level is expressed in millilitres and it will be assessed with periapical radiographs taken pre-extraction and 24-week post augmentation.
Presence of bone around the alveolar ridge Concentration (in nanograms) of gene expression for bone markers | Outcome data will be obtained at week 24
  The presence of bone around the alveolar ridge will be assessed using histology (qualitative assessment of bone infiltration)
  A Polymerase Chain Reaction (PCR) test will be done to determine the concentration (in nanograms) of gene expression for bone markers (including osteopontin, osteocalcin) at 24-week post augmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Ihtesham Rehman, PhD, Study Chair — University of Central Lancashire
Locations (6):
- United Kingdom (6):
  - University of Central Lanchashire, Preston, Lancashire
  - Devonshire House Dental Practice, Cambridge
  - St Faith's Dental Clinic,, East Grinstead
  - Halesowen Dental, Halesowen
  - Imperical College,London, London
  - UCLan community Dentists, Preston

IPD SHARING:
Plan to Share IPD: Yes
All data obtained from each participant will be anonymised at their last dental visit and any identifiable paper records, except consent forms, will be securely destroyed. The fully anonymised data set will be available in perpetuity to other researchers in the UCLanData OA repository under the open data policy.
Supporting Information: Study Protocol, SAP
Time Frame: According to UCLan's Research Data Management Policy, all digital research data that has been selected by the Data Steward or research group for retention should be deposited in the UCLan data repository or a suitable national or international data service or subject repository within 12 months of generation.
  The fully anonymised data set will be available in perpetuity to other researchers in the UCLanData OA repository under the open data policy.
Access Criteria: When the data is deposited at the UCLanData OA repository, a digital object identifier (DOI) which is unique to the dataset and ensures it continues to be accessible will be created. The DOI for the data collected in this research will be provided in the research publication.

REFERENCES:
- [Background] Solakoglu O, Gotz W, Heydecke G, Schwarzenbach H. Histological and immunohistochemical comparison of two different allogeneic bone grafting materials for alveolar ridge reconstruction: A prospective randomized trial in humans. Clin Implant Dent Relat Res. 2019 Oct;21(5):1002-1016. doi: 10.1111/cid.12824. Epub 2019 Aug 19. PMID 31424173
- [Background] Rignon-Bret C, Hadida A, Aidan A, Nguyen TH, Pasquet G, Fron-Chabouis H, Wulfman C. Efficacy of bone substitute material in preserving volume when placing a maxillary immediate complete denture: study protocol for the PANORAMIX randomized controlled trial. Trials. 2016 May 20;17(1):255. doi: 10.1186/s13063-016-1380-7. PMID 27206923

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT05938114/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT05938114/ICF_001.pdf